CLINICAL TRIAL: NCT01132014
Title: A Pilot Clinical Trial of Dendritic Cell Vaccine Loaded With Autologous Tumor for Recurrent Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Autologous OC-DC Vaccine in Ovarian Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 19809
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-04

CONDITIONS: Chemotherapy; Tumor; Ovarian Cancer
Keywords: Subjects with recurrent ovarian, fallopian tube or primary peritoneal cancer,; from whom solid tumor or ascites have been harvested and are available and; sufficient for tumorlysate preparation;and whose largest tumor nodule is 4.5; cm. Subjects may have undergone chemotherapy or other therapy following; tumor harvesting and prior to enrollment.
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

INTERVENTIONS:
Biological: OCDC — OCDC,an autologous vaccine comprised of autologous dendritic cells (DC) loaded in vitro with lysate from autologous oxidized tumor cells, administered intranodally alone, or in combination with either intravenous Daclizumab, or with a combination of Daclizumab and intravenous Bevacizumab.

SUMMARY:
This is a Five cohort sequential clinical trial for subjects with recurrent ovarian, fallopian tube, or primary peritoneal cancer to determine the feasibility and safety as well as immunogenicity of OC-DC, an autologous vaccine comprised of autologous dendritic cells (DC) loaded in vitro with lysate from autologous oxidized tumor cells, administered intranodally alone, or in combination with intravenous Bevacizumab and cyclophosphamide or in combination with intravenous Bevacizumab, cyclophosphamide and aspirin. Study duration is 24 months.

ELIGIBILITY:
Inclusion Criteria Subject has recurrent ovarian (including low malignant potential), fallopian tube, or primary peritoneal cancer.

* Subject has had prior cytoreductive surgery yielding tumor for lysate preparation.
* Lysate must meet release criteria
* Subject is 18 years of age or older.
* Subject has an ECOG performance status of less than or equal to 1.
* Subject must understand and sign the study specific informed consent.
* Subject may have received chemotherapy or other therapy after harvest of tumor and prior to enrollment. Subjects who have achieved complete response following chemotherapy are still eligible for participation
* Subject is platinum-sensitive (progression-free interval ≥ 6 months prior to recent recurrence) or platinum-resistant (progression-free interval < 6 months prior to recent recurrence).
* Subject has recovered from toxicities of prior chemotherapy or other therapy (to grade 2 or less).
* Subject may have received prior investigational therapy (including immune therapy).
* Subject may have received prior hormonal therapy.
* Subject may have received prior radiation therapy (except to inguinal region) but must have completed such therapy prior to enrollment.
* Subject has had at least 4 weeks of postoperative recovery from surgery prior to enrollment to ensure complete wound healing. Subjects with bowel resections at surgery who enroll in cohort 2 will begin protocol at least 42 days after surgery if debulking surgery had comprised of bowel resection or other bowel surgery.
* Subjects who screen fails can be re-enrolled if the causation of the screen fail has been corrected.

EXCLUSION CRITERIA

* Subject for whom tumor lysate does not meet release criteria
* Subject has a positive serum Yo antibody
* Subject whose groins are not accessible.
* Subject has a chronic or acute hepatitis C infection. Subject with an old infection that has cleared may be included.
* Subject has a chronic or acute hepatitis B infection. Subject with an old infection that has cleared may be included.
* Subject has positive test result at the screening visit for one or more of the following:

  1. HTLV-1/2
  2. Anti-HIV 1 Antibody (α-HIV-1)
* Subject requires or is likely to require more than a two-week course of corticosteroids for intercurrent illness. Subject must complete the course of corticosteroids 2 weeks before screening to meet eligibility.
* Subject has renal insufficiency as defined by a serum creatinine greater than 2.2 mg/dl or BUN greater than 40 mg/dl. Note: If creatinine is greater than 1.5 x ULN, creatinine clearance must be greater than 60ml/min.
* Subject has proteinuria greater than 3.5 gm over 24 hrs are not eligible for the study (cohort 2 only)
* Subject with liver failure as defined by a serum total bilirubin greater than 2.0 and/or serum transaminases greater than 3X the upper limits of normal.
* Subject has hematopoietic failure at baseline as defined by one of the following:

  1. Platelets less than 100,000/ mm3
  2. WBC less than 2,500/mm3
  3. Absolute Neutrophil Count (ANC) less than 1,000/mm3
  4. Absolute lymphocyte count less than 200/ mm3
  5. Hematocrit less than or equal to 30 percent
* Subject has any acute infection that requires specific therapy. Acute therapy must have been completed within seven days prior to study enrollment.
* Subject has a serious, non-healing wound, ulcer, or bone fracture.
* Subject has a clinically significant cardiovascular disease including:
* Uncontrolled hypertension;
* Myocardial infarction or unstable angina within 6 months prior to enrollment
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Subject has a grade II or greater peripheral vascular disease.
* Subject has a clinically significant peripheral artery disease, e.g., those with claudication, within 6 months.
* Subject has any underlying conditions, which would contraindicate therapy with study treatment (or allergies to reagents used in this study).
* Subject has organ allografts.
* Subject is receiving medication(s) that might affect immune function. Use of H2 antagonists are prohibited as are all antihistamines five days before and five days after each injection of study vaccine. However, NSAIDS including COX-2 inhibitors, acetaminophen or aspirin are permitted.
* Subject has clinical symptoms or signs of partial or complete gastrointestinal obstruction or who require parenteral hydration and/or nutrition (For cohort 2, 3, 4 and 5).
* Subjects with a History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess.
* Subjects with evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-05; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Safety | 30 days of last vaccination
  Safety will be established by grading the observed toxicities using the NCI Common Toxicity Criteria (CTC Version3.0). All toxicities observed within 30 days of last vaccination will be included.

SECONDARY OUTCOMES:
Clinical Response
  Clinical Response will be determined by RECIST criteria. Response rate is the proportion of patients that achieve CR or PR.
Dose limiting toxicity
  Dose-limiting toxicity is defined as: any Grade 3 or higher allergic, autoimmune or injection site reaction or any Grade 4 hematologic or non-hematologic toxicity (except fever).
Immune Response Immune Response
  Immune response will be evaluated by IFN-g ELISPOT analysis of tumor-reactive T cells, and in HLAA2+ subjects, by tetramer analysis of Her-2 specific T cells in peripheral blood. Response is defined by a 3 fold increase relative to pre-vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Ovarian Cancer Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chiang CL, Maier DA, Kandalaft LE, Brennan AL, Lanitis E, Ye Q, Levine BL, Czerniecki BJ, Powell DJ Jr, Coukos G. Optimizing parameters for clinical-scale production of high IL-12 secreting dendritic cells pulsed with oxidized whole tumor cell lysate. J Transl Med. 2011 Nov 14;9:198. doi: 10.1186/1479-5876-9-198. PMID 22082029